CLINICAL TRIAL: NCT03417284
Title: Prospective Phase I/II Trial to Jointly Optimize the Administration Schedule(s) and Dose(s) of Melphalan for Injection (Evomela) as a Preparative Regimen for Autologous Hematopoietic Stem Cell Transplantation in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Melphalan Hydrochloride in Treating Participants With Newly-Diagnosed Multiple Myeloma Undergoing Donor Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0399; NCI-2018-00906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0399 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-07

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (melphalan hydrochloride, HSCT, filgrastim) (Experimental): PREPARATIVE REGIMEN: Participants receive melphalan hydrochloride IV over 30-60 minutes on day -2.
  TRANSPLANT: Participants in both groups undergo donor stem cell transplantation IV on day 0 over 30-60 minutes.
  POST-TRANSPLANT: Participants in both groups receive filgrastim-sndz SC QD starting on day 5 and continuing in the absence of disease progression, unacceptable toxicity, or until evidence of an ANC of 0.5 x 10^9/L.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Filgrastim-sndz; Drug: Melphalan Hydrochloride
- Group 2 (melphalan hydrochloride, HSCT, filgrastim) (Experimental): PREPARATIVE REGIMEN: Participants receive melphalan hydrochloride IV over 8-9 hours on day -2.
  TRANSPLANT: Participants in both groups undergo donor stem cell transplantation IV on day 0 over 30-60 minutes.
  POST-TRANSPLANT: Participants in both groups receive filgrastim-sndz SC QD starting on day 5 and continuing in the absence of disease progression, unacceptable toxicity, or until evidence of an ANC of 0.5 x 10^9/L.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Filgrastim-sndz; Drug: Melphalan Hydrochloride

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: AHSCT; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Melphalan Hydrochloride — Given IV
  Other Names: Alkeran; Alkerana; Evomela

SUMMARY:
This phase I/II trial studies the side effects and best dose of melphalan hydrochloride in treating participants with newly-diagnosed multiple myeloma who are undergoing a donor stem cell transplantation. Giving chemotherapy before a donor stem cell transplantation helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the participant, they may help the participant's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving melphalan hydrochloride before a donor stem cell transplantation may work better than standard chemotherapy in helping to prevent multiple myeloma from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the optimal dose and schedule of melphalan for injection (melphalan hydrochloride [Evomela]) prior to autologous hematopoietic stem cell transplantation (auto-HCT) for multiple myeloma (MM).

II. To collect the pharmacokinetic data and compare the exposure-response evaluations between the 2 infusion schedules.

SECONDARY OBJECTIVES:

I. To determine the incidence of treatment related mortality (TRM) at day 90 after auto-HCT in newly diagnosed myeloma patients treated on different schedules and doses of Evomela.

II. To determine the rate of minimal residual disease (MRD) negative complete response (CR) rate at day 90 after auto-HCT in newly diagnosed myeloma patients treated on different schedules and doses of Evomela.

III. To determine the progression-free survival (PFS) after auto-HCT in newly diagnosed myeloma patients treated on different schedules and doses of Evomela.

OUTLINE: This is a phase I, dose escalation study of melphalan hydrochloride followed by a phase II study.

PREPARATIVE REGIMEN: Participants are randomized to 1 of 2 groups.

GROUP 1: Participants receive melphalan hydrochloride intravenously (IV) over 30-60 minutes on day -2.

GROUP 2: Participants receive melphalan hydrochloride IV over 8-9 hours on day -2.

TRANSPLANT: Participants in both groups undergo donor stem cell transplantation IV on day 0 over 30-60 minutes.

POST-TRANSPLANT: Participants in both groups receive filgrastim-sndz subcutaneously (SC) once daily (QD) starting on day 5 and continuing in the absence of disease progression, unacceptable toxicity, or until evidence of an absolute neutrophil count (ANC) of 0.5 x 10^9/L.

After completion of study treatment, participants are followed up at 3 months, every 3 months for 1 year, and then annually for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-relapsed multiple myeloma in complete response (CR), partial remission (PR), very good partial remission (VGPR), or symptomatic stable disease (no evidence of progression) including patients with light chain multiple myeloma (MM) detected in the serum by free light chain assay OR
* Patients with non-secretory multiple myeloma (absence of a monoclonal protein [M protein] in serum as measured by electrophoresis [serum protein electrophoresis (SPEP)] and immunofixation (serum immunofixation electrophoresis [SIFE]) and the absence of Bence Jones protein in the urine [urine protein electrophoresis (UPEP)] defined by use of conventional electrophoresis and immunofixation [urine immunofixation electrophoresis (UIFE) techniques]) but with measurable disease on imaging studies like magnetic resonance imaging (MRI), computed tomography (CT) scan or positron emission tomography (PET) scan.
* Patients who have received at least two cycles of initial systemic therapy and are within 2 to 12 months of the first dose. Mobilization therapy is not considered initial therapy.
* Karnofsky performance score 70% or higher.
* Left ventricular ejection fraction at rest > 40% within 3 months of registration.
* Bilirubin < 2 x the upper limit of normal (except patients with Gilbert syndrome in whom bilirubin level of > 2 x upper normal limit will be allowed)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x the upper limit of normal.
* Creatinine clearance of >= 40 mL/min, estimated or calculated using the Cockcroft-Gault equation.
* Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), forced vital capacity (FVC) > 50% of predicted value (corrected for hemoglobin) within 3 months of registration.
* All female and male subjects of reproductive potential must consent to the use of effective contraceptive methods as advised by the study doctor during treatment.
* Signed informed consent form.

Exclusion Criteria:

* Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms).
* Patients seropositive for the human immunodeficiency virus (HIV).
* Patients with history of myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patients participating in an investigational new drug protocol within 14 days before enrollment.
* Female patients who are pregnant (positive beta-human chorionic gonadotropin [b-HCG]) or breast feeding.
* Prior hematopoietic cell transplantation allogeneic or autologous (A prior autologous HCT will be allowed as long as it was part of tandem transplantation).
* Prior organ transplant requiring immunosuppressive therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qaiser Bashir, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered in MD Anderson Cancer Center.
Groups:
- Group1_Dose 1 200mgm2; Group 1_Dose 2 225mgm2: PREPARATIVE REGIMEN: Participants receive melphalan IV over 30-60 minutes on day -2.
  TRANSPLANT: Participants in both groups undergo donor stem cell transplantation IV on day 0 over 30-60 minutes.
  POST-TRANSPLANT: Participants in both groups receive filgrastim-sndz SC QD starting on day 5 and continuing in the absence of disease progression, unacceptable toxicity, or until evidence of an ANC of 0.5 x 10^9/L.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo HSCT
  Filgrastim-sndz: Given SC
  Melphalan Hydrochloride: Given IV
- Group 2_Dose 1 200mgm2; Group 2_Dose 225mgm2: PREPARATIVE REGIMEN: Participants receive melphalan IV over 8-9 hours on day -2.
  TRANSPLANT: Participants in both groups undergo donor stem cell transplantation IV on day 0 over 30-60 minutes.
  POST-TRANSPLANT: Participants in both groups receive filgrastim-sndz SC QD starting on day 5 and continuing in the absence of disease progression, unacceptable toxicity, or until evidence of an ANC of 0.5 x 10^9/L.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo HSCT
  Filgrastim-sndz: Given SC
  Melphalan Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
Started | 4 | 27 | 4 | 27
Completed | 3 | 27 | 3 | 27
Not Completed | 1 | 0 | 1 | 0
Not completed — Inadequate supply on study drug | 1 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2 | Total
Number analyzed (Participants) | 4 | 27 | 4 | 27 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 19 | 4 | 22 | 47
  >=65 years | 2 | 8 | 0 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 12 | 2 | 5 | 20
  Male | 3 | 15 | 2 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 4 | 9
  Not Hispanic or Latino | 3 | 24 | 3 | 23 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 27 | 4 | 27 | 62

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose and Schedule of Evomela Prior to Autologous Transplant.
Description: Dose limiting toxicity will be defined as grade 4 mucositis or any grade 4 or 5 non-hematologic or non-infectious toxicity occurring within 30 days from the start of infusion.
Time Frame: Within 30 days after the start of infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
Number analyzed (Participants) | 4 | 27 | 4 | 27
Participants
  Grade 4 Mucositis | 0 | 0 | 0 | 0
  Grade 4 non-hematologic or non-infectious toxicity | 0 | 0 | 0 | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Number of participants that are still alive and disease free one year post autologous transplant.
Time Frame: From the date of Evomela injection up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
Number analyzed (Participants) | 4 | 27 | 4 | 27
Participants | 2 | 21 | 2 | 21

3. Secondary Outcome: Treatment Related Mortality (TRM).
Description: Number of participants expired from non-disease relapse within 90 days post transplant
Time Frame: At day 90 post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
Number analyzed (Participants) | 4 | 27 | 4 | 27
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants That Have Achieved Complete Response (CR).
Description: Number of participants that have achieved Complete response (CR). Complete response definition is negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow aspirates.
Time Frame: At 90 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
Number analyzed (Participants) | 4 | 27 | 4 | 27
Participants | 1 | 13 | 2 | 13

ADVERSE EVENTS:
Time Frame: Up to one year
Arm/Group | Group1_Dose 1 200mgm2 | Group 1_Dose 2 225mgm2 | Group 2_Dose 1 200mgm2 | Group 2_Dose 225mgm2
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/27 | 0/4 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/27 | 0/4 | 0/27
Other Adverse Events (participants affected / at risk) | 3/4 | 27/27 | 4/4 | 27/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group1_Dose 1 200mgm2 (N=4) | Group 1_Dose 2 225mgm2 (N=27) | Group 2_Dose 1 200mgm2 (N=4) | Group 2_Dose 225mgm2 (N=27)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (8) | 1 (1) | 8 (8)
ALK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ALT increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
AST increased (Investigations) | 0 (0) | 5 (5) | 0 (0) | 5 (5)
Bacterial (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 25 (25) | 3 (3) | 25 (25)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dysrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Engraftment syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 9 (9) | 1 (1) | 13 (13)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fluid overload (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 27 (27) | 4 (4) | 27 (27)
Oral mucositis (Gastrointestinal disorders) | 2 (2) | 17 (17) | 3 (3) | 13 (13)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
T bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03417284/Prot_SAP_000.pdf